CLINICAL TRIAL: NCT00852540
Title: A Randomized, Double-Blind, Double Dummy, Comparative, Multicenter Study to Assess the Safety and Efficacy of Topical Retapamulin Ointment, 1%, Versus Oral Linezolid in the Treatment of Secondarily-Infected Traumatic Lesions and Impetigo Due to Methicillin-Resistant Staphylococcus Aureus
Brief Title: Retapamulin Versus Linezolid in the Treatment of SITL and Impetigo Due to MRSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110978
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Skin Infections, Bacterial
Keywords: impetigo; methicillin-resistant Staphylococcus aureus; linezolid; secondarily-infected traumatic lesion; uncomplicated skin infection; retapamulin
MeSH Terms: conditions — Cellulitis; Impetigo | interventions — Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Retapamulin (Experimental)
  Interventions: Drug: Retpamulin Ointment, 1%
- Linezolid (Active Comparator)
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Retpamulin Ointment, 1% — Topical retapamulin (SB-275833) ointment, 1% (w/w), and placebo ointment, will be provided as approximately 10 grams of an off-white smooth ointment in collapsible aluminum tubes with reverse-taper puncture-tip caps. Retapamulin or placebo ointment will be applied twice daily for 5 days.
  Arms: Retapamulin
Drug: Linezolid — Adult and adolescent (=>12 years of age) subjects will receive one 600mg linezolid tablet (overencapsulated), or one placebo capsule, twice daily for 10 days. Pediatric subjects aged 5-11 years will receive 10mg/kg body weight of a 100mg/5mL oral linezolid suspension, or placebo suspension, twice daily for 10 days. Pediatric subjects <5 years of age will receive 10mg/kg of a 100mg/5mL oral linezolid suspension, or placebo suspension, three times daily for 10 days.
  Arms: Linezolid

SUMMARY:
The purpose of this study is to provide further evidence of the clinical and bacteriological efficacy of retapamulin in the treatment of subjects with SITL or impetigo due to MRSA. Subjects aged 2 months and older will be treated with either topical retapamulin for 5 days or oral linezolid for 10 days. The primary endpoint is the clinical response at follow-up (7-9 days after the end of therapy) in subjects who have a MRSA infection at baseline. The primary population is the per-protocol MRSA population. It is anticipated that approximately 500 subjects may be enrolled in order to obtain approximately 105 subjects who have a baseline MRSA infection.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, double dummy, multicenter, comparative study in subjects 2 months of age and older with SITL (including secondarily-infected lacerations, sutured wounds and abrasions) or impetigo (bullous and non-bullous) due to MRSA. A laceration or sutured wound cannot exceed 10 cm in length with surrounding erythema not extending more than 2 cm from the edge of the lesion. Abrasions cannot exceed 100 cm2 in total area, or up to a maximum of 2% total body surface area for subjects <18 years of age, with surrounding erythema not extending more than 2 cm from the edge of the abrasion. Subjects with impetigo can have up to 10 lesions and the infected lesion(s) must not be more than 100 cm2 in area (or up to a maximum of 2% total body surface area for subjects <18 years of age), must not require surgical intervention and must be able to be appropriately treated with a topical antibiotic.

There are five study visits occurring over a 17-19 day period. At the baseline visit (Visit 1, day 1), subjects will be randomized to receive retapamulin (plus oral placebo) or linezolid (plus placebo ointment) in a 2:1 ratio. Retapamulin is applied twice daily for 5 days, and linezolid is dosed, depending on subject age, either twice or three times daily for 10 days. The on-therapy, end of therapy and follow-up visits are staggered due to the difference in duration of the treatment regimens. Subjects will be monitored and clinically evaluated at all postbaseline visits.

Randomization will be center-based and stratified by age (<5 years, ≥5 to <12 years, ≥12 years), performed using an appropriate Interactive Voice Response System (IVRS), an automated telephone system. The block size will remain confidential. Subjects are considered to have completed the study if they meet all inclusion/exclusion criteria, are considered compliant with study medication, and attend all study visits as defined by the protocol.

ELIGIBILITY:
Inclusion Criteria:

* 2 months of age or older
* diagnosis of secondarily-infected traumatic lesion (SITL) or impetigo (bullous or non-bullous)
* negative urine pregnancy test (females of childbearing potential)
* total skin infection rating scale (SIRS) score of at least 8, which must include a pus/exudate score of at least 3
* subject or parent/legal guardian willing and able to comply with protocol
* written informed, dated consent, and written assent (if applicable)

Exclusion Criteria:

* previous hypersensitivity to pleuromutilins or oxazolidinones
* phenylketonuria or known hypersensitivity to aspartame
* secondarily-infected animal/human bite, or puncture wound
* abscess
* chronic ulcerative lesion
* underlying skin disease (eg, eczematous dermatitis) with secondary infection
* systemic signs and symptoms of infection
* skin infection not appropriate for treatment by a topical antibiotic (eg, extensive cellulitis, furunculosis)
* subject requires surgical intervention for infection prior to study or likely will during the study
* receipt of systemic antibacterial or steroid, or application of any topical therapeutic agent directly to wound within 24 hours of entry into the study
* subject currently receiving adrenergic agents
* subject currently receiving serotonergic agents
* history of pseudomembranous colitis
* known, pre-existing myelosuppression, history of myelosuppression with linezolid use, or receiving a medication that produces bone marrow suppression
* history of siezures
* history of severe renal failure and undergoing dialysis
* serious underlying disease that could be imminently life-threatening
* pregnant, breast feeding or planning a pregnancy, or not using accepted method of contraception (females of childbearing potential or <1 year post-menopausal)
* use of another investigational drug within 30 days prior to entry into this study
* previously enrolled in this study
* fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency (for subjects <12 years of age receiving linezolid suspension)

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (49):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Bentonville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Paragould, Arkansas
  - GSK Investigational Site, Bakerfield, California
  - GSK Investigational Site, Bell Gardens, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Atlantis, Florida
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Grand Blanc, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Carlisle, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Hazleton, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Duncanville, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tanus T, Scangarella-Oman NE, Dalessandro M, Li G, Breton JJ, Tomayko JF. A randomized, double-blind, comparative study to assess the safety and efficacy of topical retapamulin ointment 1% versus oral linezolid in the treatment of secondarily infected traumatic lesions and impetigo due to methicillin-resistant Staphylococcus aureus. Adv Skin Wound Care. 2014 Dec;27(12):548-59. doi: 10.1097/01.ASW.0000456631.20389.ae. PMID 25396674
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 110978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110978 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo: Retapamulin ointment was administered topically twice daily (BID) for 5 days. The ointment formulation was to be applied to the infected lesion(s) at a dose of approximately 10 milligrams (mg) per centimeter squared (cm^2). Placebo was to be dosed, depending on participant age, either BID or three times a day (TID) for 10 days. Placebo oral suspension and oral tablet were formulated to appear identical to the linezolid formulations. Adolescent and adult participants (>=12 years of age) were dosed BID with 600 mg placebo tablets, pediatric participants 5 to 11 years of age were dosed with oral suspension at 0.5 milliliters (ml)/kilogram (kg) BID, and pediatric participants less than 5 years of age were dosed with oral suspension at 0.5 ml/kg TID.
- Linezolid Plus Placebo Ointment: Linezolid was to be dosed, depending on participant age, either BID or TID for 10 days. Adolescent and adult participants (>=12 years of age) were dosed BID with 600 mg tablets for 10 days. Pediatric participants who were 5-11 years of age were dosed with a 100 mg/5 ml oral suspension at a dose of 10 mg/kg BID for 10 days. Pediatric participants who were <5 years of age were dosed with a 100 mg/5 ml oral suspension at a dose of 10 mg/kg TID for 10 days. Placebo ointment was administered topically BID for 5 days.
Period: Overall Study
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Started | 270 | 140
Completed | 234 | 122
Not Completed | 36 | 18
Not completed — Adverse Event | 10 | 3
Not completed — Lack of Efficacy | 15 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 2 | 3
Not completed — Investigator Discretion | 2 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Did Not Receive Study Drug | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment | Total
Number analyzed (Participants) | 267 | 137 | 404
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characterisitcs were collected in all participants in the Intent-to-Treat Clinical (ITTC) Popluation, comprised of all randomized participants who took at least one dose of study medication. Three participants in both treatment groups were randomized but did not receive study medication.
  Years | 34.6 (21.37) | 33.8 (22.38) | 34.3 (21.69)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characterisitcs were collected in all participants in the Intent-to-Treat Clinical (ITTC) Popluation, comprised of all randomized participants who took at least one dose of study medication. Three participants in both treatment groups were randomized but did not receive study medication.
  Participants
    Female | 108 | 49 | 157
    Male | 159 | 88 | 247
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characterisitcs were collected in all participants in the Intent-to-Treat Clinical (ITTC) Popluation, comprised of all randomized participants who took at least one dose of study medication. Three participants in both treatment groups were randomized but did not receive study medication.
  participants
    African American/African Heritage | 16 | 10 | 26
    American Indian or Alaska Native | 5 | 0 | 5
    Central/South Asian Heritage | 1 | 1 | 2
    East Asian Heritage | 0 | 1 | 1
    Japanese Heritage | 5 | 2 | 7
    South East Asian Heritage | 3 | 0 | 3
    Native Hawaiian or other Pacific Islander | 5 | 1 | 6
    Arabic/North African Heritage | 0 | 3 | 3
    White/Caucasian/European | 222 | 118 | 340
    White - Mixed Race | 10 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Clinical Response at Follow-up Who Had Methicillin-resistant Staphlococcus Aureus (MRSA) as a Baseline Pathogen
Description: Follow-up is defined as 7-9 days post-therapy: Day 12-14 for retapamulin; Day 17-19 for linezolid. Clinical success at follow-up was defined as the resolution of clinically meaningful signs and symptoms of infection recorded at baseline, including a pus/exudate skin infection rating scale (SIRS) score of "0." The SIRS is used by the investigator to evaluate infected lesions. Scores on the SIRS range from 0 (absent) to 6 (severe).
Time Frame: 7-9 days post-therapy; Day 12-14 for retapamulin and Day 17-19 for linezolid
Population: Intent-to-Treat MRSA (ITTMRSA) Population: all randomized participants who took at least one dose of study medication and who had an MRSA isolated at baseline.
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 72 | 38
participants | 41 | 32
Statistical Analysis 1: Comparison: Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo; Test type: Superiority or Other; percentage of participants = 56.9, 95% CI 2-sided [45.5 to 68.4] — The estimated value is the percentage of participants achieving clinical response. Confidence intervals are not adjusted for multiplicity
Statistical Analysis 2: Comparison: Linezolid Plus Placebo Ointment; Test type: Superiority or Other; Percentage of participants = 84.2, 95% CI 2-sided [72.6 to 95.8] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants Achieving Microbiological Response (MR) at Follow-up (FU) Who Had MRSA as a Baseline Pathogen (BP)
Description: MR was defined as microbiological success if, (1) for participants (par.) whose clinical outcome at end of therapy (EOT) was "clinical success (CS)/improvement," the BP was eradicated/presumed to be eradicated at EOT, or the BP was present at EOT and absent at FU, or the BP was eradicated/presumed to be eradicated at EOT, or the BP was present at EOT and par. was a "CS" such that no culture was obtained due to lack of culturable material secondary to adequate clinical response; or (2) a pathogen not previously identified at baseline was isolated at FU in a par. identified at FU as a "CS."
Time Frame: 7-9 days post-therapy; Day 12-14 for retapamulin and Day 17-19 for linezolid
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 72 | 38
participants | 41 | 32

3. Secondary Outcome: Number of Participants With Clinical Response at Follow-up
Description: as for outcome 1
Time Frame: 7-9 days post-therapy; Day 12-14 for retapamulin and Day 17-19 for linezolid
Population: Intent-to-Treat Clinical (ITTC) Population: all randomized participants (par.) who took at least one dose of study medication. One par. was randomized to retapamulin but received linezolid. This par. is summarized in the linezolid group for all baseline and safety tables, but is summarized in the retapamulin group for all efficacy tables.
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 268 | 136
participants | 161 | 112

4. Secondary Outcome: Number of Participants Who Achieved Microbiological Response (MR) at Follow-up (FU) Who Had a Baseline Pathogen (BP)
Description: as for outcome 2
Time Frame: 7-9 days post-therapy; Day 12-14 for retapamulin and Day 17-19 for linezolid
Population: Intent-to-Treat Bacteriology (ITTB) Population: all randomized participants who took at least one dose of study medication and who had a pathogen isolated at baseline.
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 177 | 78
participants | 100 | 65

5. Secondary Outcome: Number of Participants With the Indicated Clinical Outcome at the End of Therapy Who Had MRSA as a Baseline Pathogen
Description: Clinical improvement is defined as improvement of signs/symptoms of infection recorded at baseline (BL) to such an extent that no further antimicrobial therapy is necessary. Clinical failure (CF) is defined as insufficient improvement/deterioration of signs/symptoms of the infection recorded at BL, such that additional antibiotic therapy is required. Unable to determine (UTD) is defined as refusal to consent to a clinical examination, lost to follow-up. Participants who are "CF"/"Unable to Determine" at end of therapy are considered such at follow-up as well.
Time Frame: 2-4 days post-therapy; Day 7-9 for retapamulin and Day 12-14 for linezolid
Population: ITTMRSA Population
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 72 | 38
participants
  Clinical success | 20 | 28
  Clinical improvement | 42 | 9
  Clinical failure | 8 | 1
  Unable to determine | 2 | 0

6. Secondary Outcome: Number of Participants With the Indicated Microbiological Outcome at the End of Therapy Who Had MRSA as a Baseline (BL) Pathogen
Description: Eradication is the elimination of BL pathogens. Presumed eradication and presumed improvement are clinical outcomes of success or improvement, respectively, such that no culture was obtained due to lack of culturable material, secondary to adequate clinical response, and is documented in the electronic Case Report Form. Persistence is defined as BL pathogens still being present. Presumed persistence is defined as a participant that is a clinical failure with no obtained culture. "Unable to determine" was used if no determination of BL pathogen microbiological response could be made.
Time Frame: 2-4 days post-therapy; Day 7-9 for retapamulin and Day 12-14 for linezolid
Population: ITTMRSA Population
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 72 | 38
participants
  Eradication | 1 | 0
  Presumed eradication | 20 | 28
  Presumed improvement | 42 | 9
  Persistence | 4 | 1
  Presumed persistence | 4 | 0
  Unable to determine | 1 | 0

7. Secondary Outcome: Number of Participants With the Indicated Clinical Outcome at the End of Therapy
Description: as for outcome 5
Time Frame: 2-4 days post-therapy; Day 7-9 for retapamulin and Day 12-14 for linezolid
Population: ITTC Population. One par. was randomized to retapamulin but received linezolid. This par. is summarized in the linezolid group for all baseline and safety tables, but is summarized in the retapamulin group for all efficacy tables.
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 268 | 136
participants
  Clinical success | 92 | 96
  Clinical improvement | 155 | 34
  Clinical failure | 16 | 4
  Unable to determine | 5 | 2

8. Secondary Outcome: Number of Baseline Pathogens With the Indicated Microbiological Outcome at the End of Therapy
Description: as for outcome 6
Time Frame: 2-4 days post-therapy; Day 7-9 for retapamulin and Day 12-14 for linezolid
Population: ITTB Population
Measure: Number; unit: pathogens
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 177 | 78
pathogens
  Eradication | 2 | 1
  Presumed eradication | 63 | 70
  Presumed improvement | 120 | 21
  Persistence | 7 | 1
  Presumed persistence | 9 | 1
  Unable to determine | 1 | 0

9. Secondary Outcome: Number of Participants With Therapeutic Response at Follow-up
Description: Therapeutic response is defined as the combined clinical and microbiological response. Therapeutic response iss a measure of the overall efficacy response, and a therapeutic success refers to participants who had been deemed both a "clinical success" and a "microbiological success." All other combinations (other than "clinical success" + "microbiological success") were deemed failures for therapeutic response.
Time Frame: 7-9 days post-therapy; Day 12-14 for retapamulin and Day 17-19 for linezolid
Population: ITTB Population
Measure: Number; unit: participants
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 177 | 78
participants | 100 | 65

10. Secondary Outcome: Mean Scores on the Skin Infection Rating Scale at Visits 1, 2, 3, 4, and 5
Description: The investigator evaluated skin infections by grading the infected lesion for exudate (a fluid that leaks out of blood vessels into surrounding tissue)/pus, crusting, erythema (redness of the skin)/ inflammation (E/I), tissue warmth, tissue edema (swelling), itching, and pain, according to the Skin Infection Rating Scale. All parameters were graded on a scale of 0 (absent) to 6 (severe). The total score is calculated by summing the individual scores from the 7 parameters; the total score ranges from 0 to 42.
Time Frame: Visits 1 (Day 1), 2 (Day 3-4), 3 (Day 7-9), 4 (Day 12-14), and 5 (Day 17-19)
Population: ITTC Population. Only participants with non-missing Skin Infection Rating Scale scores were included in this analysis. One par. was randomized to retapamulin but received linezolid. This par. is summarized in the linezolid group for all baseline and safety tables, but is summarized in the retapamulin group for all efficacy tables.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 268 | 136
scores on a scale
  Pus/exudate, Visit 1, n=268, 136 | 3.6 (0.82) | 3.6 (0.8)
  Pus/exudate, Visit 2, n=265, 135 | 1.7 (1.37) | 1.4 (1.25)
  Pus/exudate, Visit 3, n=255, 130 | 0.6 (1.05) | 0.4 (0.74)
  Pus/exudate, Visit 4, n=237, 125 | 0.2 (0.59) | 0.1 (0.34)
  Pus/exudate, Visit 5, n=238, 122 | 0.1 (0.39) | 0.0 (0.29)
  Crusting, Visit 1, n=268, 136 | 2.2 (1.48) | 2.1 (1.49)
  Crusting, Visit 2, n=265, 135 | 1.3 (1.21) | 1.2 (1.15)
  Crusting, Visit 3, n=255, 130 | 0.9 (1.08) | 0.8 (0.91)
  Crusting, Visit 4, n=237, 125 | 0.6 (0.95) | 0.5 (0.83)
  Crusting, Visit 5, n=238, 122 | 0.3 (0.59) | 0.3 (0.73)
  E/I, Visit 1, n=268, 136 | 3.4 (1.09) | 3.4 (1.08)
  E/I, Visit 2, n=265, 135 | 2.2 (1.19) | 2.2 (1.26)
  E/I, Visit 3, n=255, 130 | 1.1 (1.15) | 1.0 (0.93)
  E/I, Visit 4, n=237, 125 | 0.5 (0.69) | 0.5 (0.73)
  E/I, Visit 5, n=238, 122 | 0.2 (0.54) | 0.2 (0.54)
  Tissue warmth, Visit 1, n=268, 136 | 2.8 (1.33) | 2.6 (1.29)
  Tissue warmth, Visit 2, n=265, 135 | 1.4 (1.22) | 1.3 (1.22)
  Tissue warmth, Visit 3, n=255, 130 | 0.6 (0.97) | 0.4 (0.69)
  Tissue warmth, Visit 4, n=237, 125 | 0.1 (0.41) | 0.1 (0.34)
  Tissue warmth, Visit 5, n=238, 122 | 0.1 (0.38) | 0.0 (0.20)
  Tissue edema, Visit 1, n=268, 136 | 2.8 (1.24) | 2.7 (1.30)
  Tissue edema, Visit 2, n=265, 135 | 1.6 (1.23) | 1.5 (1.19)
  Tissue edema, Visit 3, n=255, 130 | 0.7 (1.02) | 0.7 (0.86)
  Tissue edema, Visit 4, n=237, 125 | 0.3 (0.60) | 0.2 (0.55)
  Tissue edema, Visit 5, n=238, 122 | 0.1 (0.35) | 0.1 (0.36)
  Itching, Visit 1, n=268, 136 | 1.6 (1.51) | 1.8 (1.51)
  Itching, Visit 2, n=265, 135 | 1.0 (1.27) | 0.9 (1.11)
  Itching, Visit 3, n=255, 130 | 0.7 (1.24) | 0.6 (1.08)
  Itching, Visit 4, n=237, 125 | 0.3 (0.79) | 0.4 (0.76)
  Itching, Visit 5, n=238, 122 | 0.1 (0.42) | 0.2 (0.66)
  Pain, Visit 1, n=268, 136 | 3.2 (1.57) | 3.0 (1.65)
  Pain, Visit 2, n=265, 135 | 1.5 (1.56) | 1.2 (1.39)
  Pain, Visit 3, n=255, 130 | 0.6 (1.14) | 0.4 (0.96)
  Pain, Visit 4, n=237, 125 | 0.2 (0.60) | 0.1 (0.56)
  Pain, Visit 5, n=238, 122 | 0.1 (0.39) | 0.1 (0.45)
  Total score, Visit 1, n=268, 136 | 19.5 (5.69) | 19.2 (5.56)
  Total score, Visit 2, n=265, 135 | 10.7 (6.78) | 9.7 (6.32)
  Total score, Visit 3, n=255, 130 | 5.2 (5.83) | 4.1 (4.16)
  Total score, Visit 4, n=237, 125 | 3.6 (6.13) | 2.5 (4.13)
  Total score, Visit 5, n=238, 122 | 2.5 (6.14) | 1.6 (3.92)

11. Secondary Outcome: Mean Wound Size at Visits 1, 2, 3, 4, and 5
Description: Lesion sized was measured in centimeters squared at Visits 1, 2, 3, 4, and 5.
Time Frame: Visits 1 (Day 1), 2 (Day 3-4), 3 (Day 7-9), 4 (Day 12-14), and 5 (Day 17-19)
Population: ITTC Population. Only participants with non-missing data were included in this analysis. One par. was randomized to retapamulin but received linezolid. This par. is summarized in the linezolid group for all baseline and safety tables, but is summarized in the retapamulin group for all efficacy tables.
Measure: Mean (Standard Deviation); unit: centimeters squared (cm^2)
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Number analyzed (Participants) | 268 | 136
centimeters squared (cm^2)
  Visit 1, n=268, 136 | 7.942 (13.3124) | 5.620 (9.6215)
  Visit 2, n=265, 135 | 4.963 (8.5492) | 4.115 (9.4305)
  Visit 3, n=255, 130 | 3.270 (10.8663) | 1.776 (6.7537)
  Visit 4, n=237, 125 | 1.556 (5.2201) | 0.812 (3.4217)
  Visit 5, n=237, 122 | 0.741 (3.5977) | 0.588 (3.3623)

ADVERSE EVENTS:
Description: Serious adverse events and non-serious adverse events were collected in the Intent-to-Treat Clinical (ITTC) Popluation, comprised of all randomized participants who took at least one dose of study medication.
Arm/Group | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo | Linezolid Plus Placebo Ointment
Serious Adverse Events (participants affected / at risk) | 3/267 | 3/137
Other Adverse Events (participants affected / at risk) | 13/267 | 22/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo (N=267) | Linezolid Plus Placebo Ointment (N=137)
Cellulitis (Infections and infestations) | 2 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Retapamulin Ointment, 1% (Weight/Weight) Plus Oral Placebo (N=267) | Linezolid Plus Placebo Ointment (N=137)
Diarrhea (Gastrointestinal disorders) | 8 | 16
Nausea (Gastrointestinal disorders) | 6 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.